CLINICAL TRIAL: NCT04069208
Title: Dose-intense Idarubicin Induction in Young Patients With Acute Myeloid Leukemia
Brief Title: IA14 Induction in Young Acute Myeloid Leukemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Cao Xinxin, Associate Professor, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AML-IA14
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; ultra-high dose idarubicin; induction
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Idarubicin

STUDY DESIGN:
Intervention Model Description: Idarubicin 14mg/m2 for 3 days cytarabine 100mg/m2 every 12 hour for 7 days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IA14 (Experimental): Idarubicin 14mg/m2 for 3 days cytarabine 100mg/m2 every 12 hour for 7 days
  Interventions: Drug: Idarubicin and cytarabine induction

INTERVENTIONS:
Drug: Idarubicin and cytarabine induction — Idarubicin 14mg/m2 for 3 days cytarabine 100mg/m2 every 12 hour for 7 days

SUMMARY:
Acute myeloid leukemia (AML) is a clinically and biologically heterogeneous disease characterized by the clonal expansion of undifferentiated myeloid precursors. Although induction chemotherapy with cytarabine and daunorubicin/Idarubicin, typically called "7+3", has not changed for several decades, the best dosage of anthracycline is still unknown. Several prospective trials have demonstrated that intense dosage of anthracycline improved complete remission (CR) and overall survival (OS). Idarubicin 12mg/m2 (IA12) has been shown to be equal to dose intense daunorubicin (90 mg/m2 ) for achieving CR. Dose-intense daunorubicin 90 mg/m2 (DA90) has been shown to improve CR compared to standard dose daunorubucin 45mg/m2 in newly diagnosed AML patients. In our previous study, CR rate of induction with daunorubicin 60 mg/m2/d (3 days) and cytarabine 200 mg/m2/d days 1-7 was about 67%. Benefit of intensification seems limited to the patients without adverse cytogenetics. Wheher ultra high dose idarubicin 14mg/m2 (IA14) could further improve CR rate, give patients with adverse cytogenetics a chance to do allo-stem cell transplantation? This phase 2, prospective, single-center study is designed to evaluate the efficacy and safety of induction with idarubicin 14mg/m2/d (3 days) and cytarabine 200 mg/m2/d days 1-7 in young newly diagnosed AML patients.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, morphologically documented primary AML or AML secondary to myelodysplastic syndrome or a myeloproliferative neoplasm based on the World Health Organization (WHO) 2008 classification (at Screening)
* Must be competent and able to comprehend, sign, and date an Ethics Committee or Institutional Review Board approved Informed Consent Form (ICF) before performance of any study-specific procedures or tests;
* ≥18 yearsand ≤60 years (at Screening);
* Eastern Cooperative Oncology Group performance status 0-2 (at Screening);
* Adequate renal function defined as: Creatinine clearance rate >50 mL/min, as calculated with the modified Cockcroft Gault equation;
* Adequate hepatic function defined as: Total serum bilirubin ≤1.5 × ULN; and serum alkaline phosphatase, aspartate transaminase and alanine transaminase ≤2.5 × ULN;
* Serum electrolytes within normal limits: potassium, calcium (total or corrected for serum albumin in case of hypoalbuminemia). If outside of normal limits, subject will be eligible when electrolytes are corrected;

Exclusion Criteria:

* Diagnosis of acute promyelocytic leukemia (APL), French-American-British classification M3 or WHO classification of APL with translocation, t(15;17)(q22;q12); subjects who undergo diagnostic workup for APL and treatment with all-trans retinoic acid (ATRA), but who are found not to have APL, are eligible (treatment with ATRA must be discontinued before starting induction chemotherapy).
* Prior treatment for AML, except for the following allowances:

  1. Leukapheresis;
  2. Treatment for hyperleukocytosis with hydroxyurea;
  3. Growth factor/cytokine support;
* Uncontrolled or significant cardiovascular disease, including any of the following:

  1. Bradycardia of less than 50 beats per minute, unless the subject has a pacemaker;
  2. Diagnosis of or suspicion of long QT syndrome (including family history of long QT syndrome);
  3. Systolic blood pressure ≥180 mmHg or diastolic blood pressure ≥110 mmHg;
  4. History of clinically relevant ventricular arrhythmias (eg, ventricular tachycardia, ventricular fibrillation, or Torsade de Pointes);
  5. History of second (Mobitz II) or third degree heart block (subjects with pacemakers are eligible if they have no history of fainting or clinically relevant arrhythmias while using the pacemaker);
  6. History of uncontrolled angina pectoris or myocardial infarction within 6 months prior to Screening;
  7. History of New York Heart Association Class 3 or 4 heart failure;
  8. Complete left bundle branch block;
  9. Known history of left ventricular ejection fraction (LVEF) ≤45% or less than the institutional lower limit of normal;
* Active acute or chronic systemic fungal, bacterial, or viral infection not well controlled by antifungal, antibacterial or antiviral therapy;
* Concurrent of other malignancies, except adequately treated non-melanoma skin cancer, curatively treated in-situ disease, or other solid tumors curatively treated with no evidence of disease
* Females who are pregnant or breastfeeding;

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2019-09-03 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete remission (CR) rate | On Day 21 (window Day 21 to Day 30), a bone marrow aspirate specimen will be collected for pathology.
  the rate of patient who get CR after induction therapy

SECONDARY OUTCOMES:
Event-free survival (EFS) | Assessed up to 24 months. Event is defined as any of the following: 1)Refractory disease (or treatment failure) which is determined at the end of the Induction Phase; 2)Relapse after CR or CRi; 3)Death from any cause at any time during the study.
  EFS is defined as the duration from initiation of IA induction treatment to the date of a first event
Overall survival (OS) | OS was defined as the duration from initiation of IA induction treatment to the date of death or last follow-up assessed up to 24 months.
  OS was defined as the duration from initiation of IA induction treatment to the date of death or last follow-up
rate of Minimal Residual Disease (MRD) negativity | MRD will be tested after on Day 21 (window Day 21 to Day 30)
  Percentage of subjects achieving CR with no evidence of Minimal Residual Disease (MRD) following induction therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Li, M.D., Study Director — Peking Union Medical College Hospital
Locations (1):
- Xinxin Cao, Beijing, Beijing Municipality, China